CLINICAL TRIAL: NCT03811951
Title: Neurologic Biomarkers of Smoking Behavior
Brief Title: Neuro Biomarkers of Smoking Behavior
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Different study initiation
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ajna Hamidovic, PharmD, MS, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017-1288
Record Dates: First submitted 2018-11-09; First posted 2019-01-22 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
Keywords: Tobacco; Cigarettes; Nicotine; Insulin
MeSH Terms: conditions — Smoking Cessation; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The University of Illinois Hospital and Health Sciences System Investigational Drug Service (IDS) randomizes treatment order to study subjects and prepares drug product and placebo. All other roles, including participant, investigator, and non-IDS study personnel are masked from treatment order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): All participants receive both Novolin R (experimental drug) and 14% NaCl (Sodium Chloride) solution (placebo), to be administered in randomly assigned order on two separate testing sessions. During administration of either Novolin R or 14% NaCl, participants will receive 1 spray in each nostril every 3 minutes for a total of 6 sprays. The nasal spray bottle delivers 0.1 ml of liquid per spray. Since the concentration of insulin in Novolin R is 100 IU/mL, six sprays will deliver a 60 IU dose.
  Interventions: Drug: Novolin R
- Non-Smokers (Experimental): All participants receive both Novolin R (experimental drug) and 14% NaCl solution (placebo), to be administered in randomly assigned order on two separate testing sessions. During administration of either Novolin R or 14% NaCl, participants will receive 1 spray in each nostril every 3 minutes for a total of 6 sprays. The nasal spray bottle delivers 0.1 ml of liquid per spray. Since the concentration of insulin in Novolin R is 100 IU/mL, six sprays will deliver a 60 IU dose.
  Interventions: Drug: Novolin R

INTERVENTIONS:
Drug: Novolin R — Novolin R is a sterile, clear, aqueous, and colorless solution that contains human insulin (rDNA origin) 100 units/mL, glycerol 16 mg/mL, metacresol 3 mg/mL, zinc chloride approximately 7 mcg/mL and water for injection. The pH (potential Hydrogen) is adjusted to 7.4. Hydrochloric acid 2N (concentration) or sodium hydroxide 2N may be added to adjust pH. Novolin R vials are latex-free. The drug substance is being purchased from McKesson.
  Other Names: McKesson Corporation, Novo Nordisk

SUMMARY:
The purpose of this study is to evaluate cognition in smokers and nonsmokers. It involves administration of intranasal insulin (Novolin R), an investigational medication followed by a brief non-invasive cognitive test. All participants will receive both Novolin R and placebo in two separate testing sessions.

DETAILED DESCRIPTION:
This program of research focuses on identifying neurologic biomarkers of smoking behavior in order to develop individualized smoking cessation aids. The intranasal insulin administered is an investigational drug and has been granted IND status by the FDA (IND#129432). During the times of drug effects, the investigators will evaluate a biomarker using computerized tasks. Non-smokers and smokers will participate in two testing sessions where the biomarker will be critically evaluated after administration of intranasal insulin and compared to the cognitive processes elicited by placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-40 years
* Smokers only: Begin smoking within 5 minutes of waking (verified by carbon monoxide concentrations greater than 10 ppm).
* Non-smokers only: No self-reported cigarette use in the past 1-year period.
* Non-smokers only: Carbon monoxide concentration < 6 ppm.
* Normal vitals (blood pressure < 120/80 mmHg; heart rate between 60 and 100 bpm, body temperature <37 °C)
* Point-of-care (POC) blood glucose between 80 and 140 mg/dL
* Body mass index between 18.5 and 30 kg/m2

Exclusion Criteria:

* Use of non-cigarette tobacco products, e-cigarettes, or smoking cessation treatment
* Positive urine drug screen test
* Current pregnancy (urine test-verified) or lactation, or a plan to become pregnant
* Breath Alcohol Concentration >0.00%
* Shipley IQ (Intelligence Quotient) test <80
* Hyposmic or anosmic individuals (identifying less than 10 of 12 smells correctly)
* Abnormal physical exam of the nares
* Lifetime DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) Axis 1 disorder (except anxiety and depression)
* Current DSM-5 Axis depression or anxiety disorder
* Prescription medications
* Over-the-counter psychotropic medications
* Use of any medications administered intranasally
* Allergies to any ingredients in intranasal insulin or placebo
* Braided hair that would cause noise in EEG recording

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajna Hamidovic, PharmD, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Department of Pharmacy Practice, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benowitz NL, Gourlay SG. Cardiovascular toxicity of nicotine: implications for nicotine replacement therapy. J Am Coll Cardiol. 1997 Jun;29(7):1422-31. doi: 10.1016/s0735-1097(97)00079-x. PMID 9180099
- [Background] de la Monte SM. Intranasal insulin therapy for cognitive impairment and neurodegeneration: current state of the art. Expert Opin Drug Deliv. 2013 Dec;10(12):1699-709. doi: 10.1517/17425247.2013.856877. Epub 2013 Nov 12. PMID 24215447
- [Background] Fehm HL, Perras B, Smolnik R, Kern W, Born J. Manipulating neuropeptidergic pathways in humans: a novel approach to neuropharmacology? Eur J Pharmacol. 2000 Sep 29;405(1-3):43-54. doi: 10.1016/s0014-2999(00)00540-9. PMID 11033313
- [Background] Franken IH, van Strien JW, Kuijpers I. Evidence for a deficit in the salience attribution to errors in smokers. Drug Alcohol Depend. 2010 Jan 15;106(2-3):181-5. doi: 10.1016/j.drugalcdep.2009.08.014. Epub 2009 Sep 24. PMID 19781864
- [Background] Hamidovic A, Khafaja M, Brandon V, Anderson J, Ray G, Allan AM, Burge MR. Reduction of smoking urges with intranasal insulin: a randomized, crossover, placebo-controlled clinical trial. Mol Psychiatry. 2017 Oct;22(10):1413-1421. doi: 10.1038/mp.2016.234. Epub 2017 Feb 28. PMID 28242873
- [Background] Kern W, Born J, Schreiber H, Fehm HL. Central nervous system effects of intranasally administered insulin during euglycemia in men. Diabetes. 1999 Mar;48(3):557-63. doi: 10.2337/diabetes.48.3.557. PMID 10078556
- [Background] Luijten M, van Meel CS, Franken IH. Diminished error processing in smokers during smoking cue exposure. Pharmacol Biochem Behav. 2011 Jan;97(3):514-20. doi: 10.1016/j.pbb.2010.10.012. Epub 2010 Oct 31. PMID 21047524
- [Background] Nedelcovych MT, Gadiano AJ, Wu Y, Manning AA, Thomas AG, Khuder SS, Yoo SW, Xu J, McArthur JC, Haughey NJ, Volsky DJ, Rais R, Slusher BS. Pharmacokinetics of Intranasal versus Subcutaneous Insulin in the Mouse. ACS Chem Neurosci. 2018 Apr 18;9(4):809-816. doi: 10.1021/acschemneuro.7b00434. Epub 2018 Jan 4. PMID 29257872
- [Background] Ott V, Benedict C, Schultes B, Born J, Hallschmid M. Intranasal administration of insulin to the brain impacts cognitive function and peripheral metabolism. Diabetes Obes Metab. 2012 Mar;14(3):214-21. doi: 10.1111/j.1463-1326.2011.01490.x. Epub 2011 Nov 16. PMID 21883804
- [Background] Rass O, Fridberg DJ, O'Donnell BF. Neural correlates of performance monitoring in daily and intermittent smokers. Clin Neurophysiol. 2014 Jul;125(7):1417-26. doi: 10.1016/j.clinph.2013.12.001. Epub 2013 Dec 11. PMID 24380760
- [Background] Reger MA, Craft S. Intranasal insulin administration: a method for dissociating central and peripheral effects of insulin. Drugs Today (Barc). 2006 Nov;42(11):729-39. doi: 10.1358/dot.2006.42.11.1007675. PMID 17171192
- [Background] Schmid V, Kullmann S, Gfrorer W, Hund V, Hallschmid M, Lipp HP, Haring HU, Preissl H, Fritsche A, Heni M. Safety of intranasal human insulin: A review. Diabetes Obes Metab. 2018 Jul;20(7):1563-1577. doi: 10.1111/dom.13279. Epub 2018 Apr 6. PMID 29508509
- [Background] Shemesh E, Rudich A, Harman-Boehm I, Cukierman-Yaffe T. Effect of intranasal insulin on cognitive function: a systematic review. J Clin Endocrinol Metab. 2012 Feb;97(2):366-76. doi: 10.1210/jc.2011-1802. Epub 2011 Dec 7. PMID 22162476
- [Background] Strachan MW. Insulin and cognitive function in humans: experimental data and therapeutic considerations. Biochem Soc Trans. 2005 Nov;33(Pt 5):1037-40. doi: 10.1042/BST20051037. PMID 16246040
- [Background] West R, Hajek P, Foulds J, Nilsson F, May S, Meadows A. A comparison of the abuse liability and dependence potential of nicotine patch, gum, spray and inhaler. Psychopharmacology (Berl). 2000 Apr;149(3):198-202. doi: 10.1007/s002130000382. PMID 10823399

RESULTS

PARTICIPANT FLOW:
Groups:
- Novolin R First, Then Placebo: Participants received active ingredients of intranasal insulin, Novolin R, every 3 minutes for the total of 6 sprays in session 1. Then, participants received placebo intranasal spray every 3 minutes for the total of 6 sprays in session 2.
- Placebo First, Then Novolin R: Participants received placebo intranasal spray every 3 minutes for the total of 6 sprays in session 1. Then, participants received active ingredients of intranasal insulin, Novolin R, every 3 minutes for the total of 6 sprays in session 2.
Period: First Intervention (1 Day)
Arm/Group | Novolin R First, Then Placebo | Placebo First, Then Novolin R
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Novolin R First, Then Placebo | Placebo First, Then Novolin R
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Novolin R First, Then Placebo | Placebo First, Then Novolin R
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novolin R First, Then Placebo | Placebo First, Then Novolin R | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 24 [21 to 27] | 24.5 [21 to 28] | 24.25 [21 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  American Indian/Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown/do not want to specify | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Go/No-Go Accuracy
Description: Go/No-Go is used to measure a participants capacity for sustained attention and response control. The test requires a participant to perform an action given certain stimuli (e.g., press a button - Go) and inhibit that action under a different set of stimuli (e.g., not press that same button - No-Go).
  Average of the 2 runs (run 1 - insulin; run 2 - placebo) were calculated for mean reaction time (+SEM) of smokers and non-smokers on no-go stimuli. The minimum reaction time was 23.08 ms and the maximum reaction time was 97.44 ms. The higher mean value represents slower the reaction time, and the lower mean value represents quicker the reaction time. The higher value means that participants have difficulties with inhibiting a prepotent response. The values do not represent a better or worse outcome.
Time Frame: From time of drug administration to 70 minutes following drug administration, up to 90 minutes
Population: All the participants were non-smokers
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Smokers | Non-Smokers
Number analyzed (Participants) | 0 | 4
Milliseconds
  Run 1 (Insulin) |  | 70.771 (25.82)
  Run 2 (Placebo) |  | 67.693 (27.95)

ADVERSE EVENTS:
Time Frame: 2 sessions, up to 2 days
Description: All-Cause Mortality and Serious Adverse Events were monitored/assessed, but none observed
Groups:
- Novolin R (First Intervention): Participants received active ingredients of intranasal insulin, Novolin R, every 3 minutes for the total of 6 sprays in first session.
- Placebo (First Intervention): Participants received placebo intranasal spray every 3 minutes for the total of 6 sprays in first session.
- Placebo (Second Intervention): Participants received placebo intranasal spray every 3 minutes for the total of 6 sprays in second session.
- Novolin R (Second Intervention): Participants received active ingredients of intranasal insulin, Novolin R, every 3 minutes for the total of 6 sprays in second session.
Arm/Group | Novolin R (First Intervention) | Placebo (First Intervention) | Placebo (Second Intervention) | Novolin R (Second Intervention)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Novolin R (First Intervention) (N=2) | Placebo (First Intervention) (N=2) | Placebo (Second Intervention) (N=2) | Novolin R (Second Intervention) (N=2)
Nasal Irritation (General disorders) | 2 | 1 | 1 | 1
Sweating (General disorders) | 0 | 1 | 0 | 0
Sneezing (General disorders) | 0 | 1 | 0 | 0
Decreased sense of smell, but not total loss (General disorders) | 0 | 1 | 0 | 0
Partial anosmia (blunted) (General disorders) | 1 | 0 | 0 | 0
Stinginess (General disorders) | 0 | 0 | 0 | 1
Hunger (General disorders) | 0 | 0 | 1 | 0
Dizziness (General disorders) | 0 | 0 | 1 | 0
Sinus Pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 2 | 2 | 2
Burning (General disorders) | 2 | 2 | 2 | 2
Taste (General disorders) | 2 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03811951/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03811951/Prot_SAP_001.pdf